CLINICAL TRIAL: NCT05852366
Title: Efficacy of Herbal Dentifrice for Management of Dentinal Hypersensitivity Post Scaling and Root Planning in Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Herbal Dentifrice for Management of Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Collaborators: Jasberry Healthcare Pvt. Ltd (Unknown)
Responsible Party: Principal Investigator, D. Gopalakrishnan, DEAN, Professor and HOD, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DYPV/EC/883/22
Record Dates: First submitted 2023-04-08; First posted 2023-05-10 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Dentinal Hypersensitivity; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental group): (n=25): Jasmate toothpaste preparation (Experimental): Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the Jasmate toothpaste onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 8 weeks for assessment of the efficacy
  Interventions: Drug: Toothpaste Preparation
- Group B (Positive Control): (n=25): Bioactive glass based BioMin F toothpaste preparation (Active Comparator): Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the Biomin F toothpaste (Bioactive glass with Calcium, Phosphate and Fluoride) onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 8 weeks for assessment of the efficacy
  Interventions: Drug: Toothpaste Preparation
- Group C (Negative Control): (n=25): Placebo toothpaste without any active desensitizing agent (Placebo Comparator): Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the Placebo toothpaste without any active desensitizing agent onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 8 weeks for assessment of the efficacy
  Interventions: Drug: Toothpaste Preparation

INTERVENTIONS:
Drug: Toothpaste Preparation — Dentifrice for management of dentinal hypersensitivity

SUMMARY:
* Recently, Herbal formulations have gained wide popularity in management of Dentinal hypersensitivity owing to the additive effects of active anti-inflammatory ingredients like Curcuma longa, Clove oil, Acacia arabica and Spinach leaves in addition to desensitizing ingredients like Potassium nitrate and/or Sodium fluoride.
* Jasmate herbal formulations which contains Potassium Nitrate along with aqua, calcium carbonate, sodium cocoyl glutamate, sorbitol 70%, glycerin, curcuma longa, arginine hydrochloride, erythritol, sodium saccharin, hydrated silica, sodium carboxymethyl cellulose, elettaria cardamomum, foeniculum vulgare, melaleuca leucadendra, eucalyptus globules, aloe barbadensis, carnosic acid, zinc oxide, hydroxyapatite, propolis, hippophae rhamnoides, syzygium aromaticum, myrtus communis, sodium benzoate and sodium fluoride7, where such formulations claim to have an anti-inflammatory action which further reduces the DH.
* Efficacy of desensitizing preparations containing the above ingredients, in the form of Jasmate was tested in the laboratory along with BioMin F and results were encouraging with sufficient occlusion of the dentinal tubules in both the groups without statistically significant differences in the results.
* The biocompatibility (cytotoxicity) of Jasmate toothpaste preparation was evaluated in the laboratory by using human gingival fibroblasts at different concentrations. Different tests like cell cycle analysis, apoptosis / necrosis and MTT were done and Jasmate toothpaste preparation showed the lowest cytotoxicity as compared to BioMin F toothpaste preparation. Jasmate toothpaste preparation showed more than 92% of live cells in all concentrations.
* The current randomized controlled clinical trial will be conducted to evaluate safety and efficacy of Jasmate toothpaste preparation in the management of DH post scaling and root planing in patients with chronic periodontitis.

DETAILED DESCRIPTION:
* Chronic periodontitis is an immuno-inflammatory disease characterized by inflammation of gingiva, formation of periodontal pocket, loss of attachment followed by alveolar bone destruction.
* In the presence of periodontal pocket various changes take place along the root surface (medial wall) out of which cytotoxic changes is of great importance.1
* The first approach to manage the chronic periodontitis is thorough supra-gingival and sub-gingival scaling followed by root planing to achieve clean, smooth and hard root surface.2
* One of the most common patient centered adverse outcome of scaling and root planing (Phase I therapy) is dentinal hypersensitivity which is of great clinical significance.3
* Dentinal hypersensitivity (DH) is characterized by short, sharp pain arising from exposed dentin in response to stimuli typically thermal, evaporative, tactile, osmotic, or chemical and which cannot be ascribed to any other form of dental defect or pathology.4
* DH leads to both physical and psychological issues for a patient with regards to the type of food selection, maintaining dental hygiene, and beauty aspects and also affects the quality of life.5
* There are various formulations available to manage DH both in-office and at home like potassium nitrate, potassium chloride, strontium chloride, stannous fluoride, hexahydrate, and aluminum, potassium or ferric oxalates and fluorides.6
* One of the common disadvantages of these commercially available formulations is the inadequate depth of penetration leading to partial relief from DH.
* To overcome this bioactive glass containing dentifrices (BioMin F) was introduced having stable hydroxycarbonate apatite crystal precipitaion that occludes the dentinal tubules when bioactive glass comes in contact with saliva.7 Recently, Herbal formulations have gained wide popularity in management of Dentinal hypersensitivity owing to the additive effects of active anti-inflammatory ingredients like Curcuma longa, Clove oil, Acacia arabica and Spinach leaves in addition to desensitizing ingredients like Potassium nitrate and/or Sodium fluoride.
* Jasmate herbal formulations which contains Potassium Nitrate along with aqua, calcium carbonate, sodium cocoyl glutamate, sorbitol 70%, glycerin, curcuma longa, arginine hydrochloride, erythritol, sodium saccharin, hydrated silica, sodium carboxymethyl cellulose, elettaria cardamomum, foeniculum vulgare, melaleuca leucadendra, eucalyptus globules, aloe barbadensis, carnosic acid, zinc oxide, hydroxyapatite, propolis, hippophae rhamnoides, syzygium aromaticum, myrtus communis, sodium benzoate and sodium fluoride7, where such formulations claim to have an anti-inflammatory action which further reduces the DH.
* Efficacy of desensitizing preparations containing the above ingredients, in the form of Jasmate was tested in the laboratory along with BioMin F and results were encouraging with sufficient occlusion of the dentinal tubules in both the groups without statistically significant differences in the results.
* The biocompatibility (cytotoxicity) of Jasmate toothpaste preparation was evaluated in the laboratory by using human gingival fibroblasts at different concentrations. Different tests like cell cycle analysis, apoptosis / necrosis and MTT were done and Jasmate toothpaste preparation showed the lowest cytotoxicity as compared to BioMin F toothpaste preparation. Jasmate toothpaste preparation showed more than 92% of live cells in all concentrations.
* The current randomized controlled clinical trial will be conducted to evaluate safety and efficacy of Jasmate toothpaste preparation in the management of DH post scaling and root planing in patients with chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be in good general health as determined by the Investigator/ medical expert;
* The patient should agree not to participate in any other oral/dental product studies during the course of this study;
* The patient should agree to delay any dental treatment until the study has been completed;
* The patient should agree to abstain from the use of any non-study oral hygiene products;
* The patient should exhibit adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect);
* The patient should agree to return for all scheduled visits and follow study procedures;
* The patient should have a minimum of 20 teeth
* The periodontal status of the patient should be Mild to moderate periodontitis (AAP classification 1999)
* The oral status of the patient should be as follows:

Plaque index (Silness & Löe 1964) >2 Gingival Index (Löe and Silness 1963) >1.5 Modified Sulcus Bleeding Index (Mombelli et al 1987) >1 PPD > 4mm

* The patient should have two teeth with a Schiff sensitivity score > 1 in response to air challenge.
* If these two eligible teeth are located in the same quadrant, they have to be separated by one other teeth.

Exclusion Criteria:

* Presence of any condition, abnormality or situation at baseline that in the opinion of the Principal Investigator may preclude the volunteer's ability to comply with study requirements, including completion of the study or the quality of the data
* Pregnant females
* Patients having history of Tobacco use
* Patients with Sjögren's disease
* Patients having immune deficiency diseases, i.e., HIV or AIDS
* Patients with poorly controlled diabetes mellitus
* Patients taking anti TNF-alpha medication for rheumatoid arthritis
* Patients taking anti-inflammatory, analgesic, or psychotropic drugs,
* Patients having self-reported eating disorders, uncontrolled gastroesophageal reflux disease (GERD or Acid Reflux), excessive dietary or environmental exposure to acids, or other systemic conditions that are predisposing to dentinal hypersensitivity;
* Patients with a history or presence of kidney disorders, kidney stones, celiac disease, inflammatory bowel disease (ulcerative colitis or Crohn's disease), chronic pancreatitis, have had intestinal or weight-loss surgery, or if have stomach or intestinal problems that keep them from absorbing certain foods or nutrients;
* The teeth will be excluded from study measurements if they have deep, defective, or facial restorations; have full crowns, extensive caries, cracked enamel, or are abutment teeth for fixed or removable prosthesis;
* The teeth having endo-perio lesion.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in dentinal hypersensitivity | Baseline to 8 weeks
  Dentinal hypersensitivity score will be measured by Visual analogue scores on a scale of 0 to 10 using Air stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Dharamarajan Gopalakrishnan, MDS, Ph.D, Principal Investigator — DEAN, Professor and HOD
Locations (1):
- Dr. D Y Patil dental College and Hospital, Pimpri, Pune, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No